CLINICAL TRIAL: NCT01398488
Title: Patient Education After Lung Transplantation Via Tablet Computers Versus Conventional Education - a Randomized Open Controlled Trial
Brief Title: Patient Education After Lung Transplantation Via Tablet Computers Versus Conventional Education
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hannover Medical School (Other)
Responsible Party: Principal Investigator, Thomas Fuehner, MD, Hannover Medical School
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: V 2.0 16/03/2011
Record Dates: First submitted 2011-07-05; First posted 2011-07-20 (Estimated); Last update posted 2013-06-06 (Estimated); Status verified 2013-06

CONDITIONS: Lung Transplantation
Keywords: Trough levels; Education; Adherence
MeSH Terms: interventions — Patient Education as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventional Patient education (Active Comparator): Conventional Patient education by health care professionals.
  Interventions: Behavioral: Patient education
- Patient education via Tablet computer (Experimental): Patient education after lung transplantation via Tablet computers. An electronic patient questionnaire via tablet computer will be collected in addition.
  Interventions: Behavioral: Patient education

INTERVENTIONS:
Behavioral: Patient education — Patient education by health care professional compared to education via tablet PC

SUMMARY:
Experimental intervention:

Patient education after lung transplantation via Tablet computers. An electronic patient questionnaire via tablet computer will be collected in addition.

Control intervention:

Conventional Patient education by health care professionals. A paper-based patient questionnaire will be provided.

DETAILED DESCRIPTION:
Noncompliance with immunosuppressive medications after organ transplantation is thought to be a leading cause of allograft rejection, graft loss, and death. Immunosuppressant medy to prevent graft rejection after lung transplantation.

Reported non-compliance rates with calcineurin inhibitors are ranging between 13 and 22 % after lung transplantation. Incidence of non-compliance increases over time after transplantation. Increased health care costs, decreased quality of life, and organ failure (incl. the need for re-do transplantation) are possible consequences of immunosuppressant noncompliance. Therefore, medication compliance defined as the extent to which a patient's medication taking behaviour coincides with the prescribed regimen, is a critical issue in transplantation. Repeated patient education is one option to overcome non-adherence and immunosuppressive medication non-compliance.

Immunosuppressive therapy is monitored by measurement of drug levels. Fluctuating drug levels increase the risk for rejection and drug toxicities. In addition, frequent dose adjustments, case management and frequent monitoring of drug levels are cost-intensive.

ELIGIBILITY:
Inclusion Criteria:

* Patients at least 6 months after lung transplantation (single, double or combined)
* Informed consent
* At least 10 trough levels analyzed in MHH reference lab in last 6 months
* < 50% of calcineurin inhibitor trough levels in target range in last 6 months in outpatient clinic

Exclusion Criteria:

* Hospitalization during last 3 months
* BOS stage 3 (FEV1 < 50% baseline)
* End stage kidney disease (GFR <15 ml/min/1.73 m2 or renal replacement therapy)
* Oxygen requirement at rest
* Steroid pulse therapy (>500 mg methylprednisolone per day) during the last 4 weeks
* Illiteracy
* Need for isolation (Colonization with multi. or pan resistant organisms, e.g. MRSA, B. cenocepacia)
* limited German language skills or other reasons which might impair patient communication or computer handling

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2011-07; Primary Completion 2012-07 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Calcineurin trough levels | 6 month
  Improvement of percentage of calcineurin inhibitor trough levels (Delta %) in target range 6 months after patient education compared to 6 months before patient education

SECONDARY OUTCOMES:
Calcineurin trough levels variability | 6 month
  Trough level variability 6 months after patient education compared to 6 months before patient education
Interval Adherence | 6 month
  interval adherence (number of measurements vs. recommended measurements) 6 months after patient education compared to 6 months before patient education
Trough level interval | 6 month
  Interval of trough level measurement variability 6 months after patient education compared to 6 months before patient education
Total time of education | 6 month
  Total time of education
Total time of answering questionnaire | 6 month
  Total time of answering questionnaire
Knowledge Improvement | 6 month
  Improvement of patient knowledge on immunosuppressive after patient education
Self rated adherence | 6 month
  Self rated adherence to immunosuppressive medication (BAASIS scale)
Adherence | 6 month
  Therapy adherence 6 months after patient education compared to 6 months before patient education
Glomerular filtration rate | 6 month
  Glomerular filtration rate 6 months after patient education compared to baseline (CKD-EPI)

CONTACTS AND LOCATIONS:
Overall Officials: Jens T Gottlieb, MD, Principal Investigator — Hannover Medical School
Locations (1):
- Hanover Medical School, Hanover, Lower Saxony, Germany

REFERENCES:
- [Derived] Mellon L, Doyle F, Hickey A, Ward KD, de Freitas DG, McCormick PA, O'Connell O, Conlon P. Interventions for increasing immunosuppressant medication adherence in solid organ transplant recipients. Cochrane Database Syst Rev. 2022 Sep 12;9(9):CD012854. doi: 10.1002/14651858.CD012854.pub2. PMID 36094829
- [Derived] Suhling H, Rademacher J, Zinowsky I, Fuge J, Greer M, Warnecke G, Smits JM, Bertram A, Haverich A, Welte T, Gottlieb J. Conventional vs. tablet computer-based patient education following lung transplantation--a randomized controlled trial. PLoS One. 2014 Mar 7;9(6):e90828. doi: 10.1371/journal.pone.0090828. eCollection 2014. PMID 24608864